CLINICAL TRIAL: NCT05525325
Title: Mode of Sedation During Endovascular Treatment of Vertebrobasilar Stroke
Acronym: MOONRISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Dr. Silvia Schönenberger, MD, Head of Section of Neurointensive Care, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MOONRISE
Record Dates: First submitted 2022-08-23; First posted 2022-09-01 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Stroke Thrombectomy
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General Anesthesia Group (Active Comparator): Patients randomized to the GA arm are intubated after anesthetic induction.
  Interventions: Procedure: General Anesthesia
- Procedural Sedation Group (Experimental): After randomization into the PS arm, the need for analgesics or sedatives are evaluated clinically.
  Interventions: Procedure: General Anesthesia

INTERVENTIONS:
Procedure: General Anesthesia — Patients randomized to the GA arm are intubated after anesthetic induction. For this purpose, they are pre-oxygenated with an oxygen mask and non-invasive monitoring is established. After sufficient pre-oxygenation has been applied, analgesic and sedative medication are administered. If the patient is sufficiently long nil by mouth they are manually ventilated before a muscle relaxant is administered. A rapid-sequence induction is performed with administration of an opioid, sedative and muscle relaxant in rapid succession and without intermediate manual ventilation in non-nil by mouth patients. To secure the airway, an endotracheal tube is inserted into the trachea with the aid of a laryngoscope. After insertion of the endotracheal tube, its endotracheal position is confirmed with auscultation and capnography. GA maintenance therapy with opioids, sedatives and catecholamines, if needed, will then be started.

SUMMARY:
Optimal anesthetic mode is not established for patients with vertebrobasilar stroke undergoing endovascular treatment. We want to investigate whether a procedural sedation mode approach is feasible compared to general anesthesia

DETAILED DESCRIPTION:
Endovascular treatment has become standard of care for many patients with acute ischemic strokes due to large vessel occlusions and is recommended by several national and international guidelines. Several studies have shown that anesthetic modality during endovascular treatment might affect the functional outcome. While much evidence has been generated for ischemic stroke of the anterior circulation, only a few studies have investigated anesthetic modalities in strokes with occlusions of the vertebrobasilar arteries. The majority of patients with vertebrobasilar occlusion strokes undergo endovascular procedure in general anesthesia and not a less burdensome sedation despite the lack of evidence for that approach. A few retrospective studies and a small single-center prospective randomized trial investigating this topic indicate that primary procedural sedation might be a feasible anesthetic approach. Here we aim to provide further high-level evidence by conducting a prospective randomized clinical trial with a PROBE (parallel-group, open-label randomized controlled with blinded endpoint evaluation) design for this research question.

ELIGIBILITY:
Inclusion Criteria:

1. Decision for thrombectomy according to local protocol for acute recanalizing stroke treatment
2. Age 18 years or older, either sex
3. National Institutes of Health Stroke Scale (NIHSS) ≥ 4
4. Acute ischemic stroke in the posterior circulation with isolated or combined occlusion of vertebral artery (VA) and basilar artery (BA)
5. Informed consent by the patient him-/herself or his/her legal representative obtainable within 72 h of treatment (deferred consenting procedure)

Exclusion Criteria:

1. Intracerebral hemorrhage
2. Coma on admission (Glasgow Coma Scale ≤ 8)
3. Severe respiratory instability, loss of airway protective reflexes or vomiting on admission, where primary intubation and general anesthesia is deemed necessary
4. Intubated state before randomization
5. Severe hemodynamic instability (e.g. due to decompensated cardiac insufficiency)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Functional outcome as measured by modified Ranking Scale (mRS) after admission. | 90 days +/- 2 weeks
  0-6; higher mean worse outcome

SECONDARY OUTCOMES:
Early neurological improvement indicated by change of National Institute of Health Stroke Scale (NIHSS) Score 24 hours after admission | [NIHSS on admission - NIHSS after 24 hours]
  0-42 points; higher mean worse outcome
Mortality | intra-hospital until discharge up to 2 weeks [yes/no] and over the whole follow-up period up to 3 months [time to event]
  cerebral or non-cerebral cause of death
Postinterventional pc-ASPECTS, determined with CT or MRI post-interventional follow up scan | 12-36 hours after admission
  semi-quantitative method for grading irreversible ischemia in the vertebrobasilar system; 0-10 points; lower mean higher infarct volumes
Feasibility of EST | duration of thrombectomy procedure in minutes
  e.g. necessity of intubation, cardio-respiratory stability, loss in level of consciousness, loss of cough reflex, vomiting
Complications before/during and after EST | duration of the whole hospital stay in days
  e.g. severe agitation, loss of level of consciousness, loss of cough reflex, vomiting, cardio-respiratory stability

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Schönenberger, MD, Principal Investigator — University Hospital Heidelberg; Min Chen, MD, Principal Investigator — UUHeidelberg
Locations (1):
- Department of Neurology, University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jadhav AP, Bouslama M, Aghaebrahim A, Rebello LC, Starr MT, Haussen DC, Ranginani M, Whalin MK, Jovin TG, Nogueira RG. Monitored Anesthesia Care vs Intubation for Vertebrobasilar Stroke Endovascular Therapy. JAMA Neurol. 2017 Jun 1;74(6):704-709. doi: 10.1001/jamaneurol.2017.0192. PMID 28395002
- [Background] Weyland CS, Chen M, Potreck A, Jager LB, Seker F, Schonenberger S, Bendszus M, Mohlenbruch M. Sedation Mode During Endovascular Stroke Treatment in the Posterior Circulation-Is Conscious Sedation for Eligible Patients Feasible? Front Neurol. 2021 Sep 17;12:711558. doi: 10.3389/fneur.2021.711558. eCollection 2021. PMID 34603184
- [Result] Schonenberger S, Henden PL, Simonsen CZ, Uhlmann L, Klose C, Pfaff JAR, Yoo AJ, Sorensen LH, Ringleb PA, Wick W, Kieser M, Mohlenbruch MA, Rasmussen M, Rentzos A, Bosel J. Association of General Anesthesia vs Procedural Sedation With Functional Outcome Among Patients With Acute Ischemic Stroke Undergoing Thrombectomy: A Systematic Review and Meta-analysis. JAMA. 2019 Oct 1;322(13):1283-1293. doi: 10.1001/jama.2019.11455. PMID 31573636